CLINICAL TRIAL: NCT04376905
Title: Assessment of Extra Vascular Lung Water and Pulmonary Permeability by Transpulmonary Thermodilution in Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Brief Title: Extra Vascular Lung Water and Pulmonary Permeability in Critically Ill Patients With SARS-CoV-2 (COVID-19)
Acronym: PiCCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0193
Record Dates: First submitted 2020-04-16; First posted 2020-05-06 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID-19; Pneumonia; Acute Respiratory Distress Syndrome
Keywords: ARDS; ICU; Transpulmonary thermodilution; Extravascular lung water; Pulmonary Vascular Permeability Index
MeSH Terms: conditions — COVID-19; Pneumonia; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a syndromic definition of an acute lung injury with alteration of biomechanics (lower respiratory system compliance) mostly associated with increased lesional edema. Increase in Pulmonary Vascular Permeability Index (PVPI) accompanied with accumulation of excess Extravascular Lung Water (EVLW) is the hallmark of ARDS. In routine clinical practice, the investigators measure the EVLW and PVPI in ARDS patients, as suggested by expert's recommendations, using a transpulmonary thermodilution (TPTD) technique.

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a newly recognized illness that has spread rapidly throughout Wuhan (Hubei province) to other provinces in China and around the world. Most critically ill patients with SARS-CoV-2 will present the criteria for the definition of ARDS. However, many of these patients have a particular form of ARDS with severe hypoxemia often associated with near normal respiratory system compliance. This combination is almost never seen in severe ARDS. Thus other mechanisms (including probably vascular mechanisms), that are still poorly described, have to be involved in SARS-CoV-2.

EVLW and PVPI have never been assessed in SARS-CoV-2 mechanically ventilated patients. The aim of this study is to evaluate these two parameters in order to best characterize and understand the mechanisms related to SARS-CoV-2.

Based on observation of several cases in intensive care units (ICU), the investigators hypothesize that there are following different SARS-CoV-2 patterns:

1. Nearly normal compliance, low lung recruitability, normal EVLW and low PVPI.
2. Low compliance due to increased edema, high lung recruitability, high EVLW and high PVPI.

ELIGIBILITY:
Inclusion criteria:

* COVID-19 critically ill patients
* Invasive mechanical ventilation

Exclusion criteria:

* Age under 18
* Pregnancy
* Legally protected adults
* Contra-indication of using PiCCO device: jugular venous thrombosis, or severe chronic femoral/iliac artery occlusive disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Changes of Extra Vascular Lung Water | Since intubation at day 0 and measured repetitively by 6 hours until day 3
  EVLW (ml/kg) measured by a PiCCO device using TPTD thermodilution

SECONDARY OUTCOMES:
Changes of Pulmonary Vascular Permeability Index | Since intubation at day 0 and measured repetitively by 6 hours until day 3
  PVPI measured by a PiCCO device using TPTDventilation, duration of ICU length of stay, ICU mortality
Changes of pulmonary compliance | Since intubation at day 0 and measured repetitively by 6 hours until day 3
  Changes of pulmonary compliance (ml/mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Kada KLOUCHE, MD PhD, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC